CLINICAL TRIAL: NCT02333890
Title: A Phase 2 Randomized, Double-blind, Window of Opportunity Trial Evaluating Clinical and Correlative Effects of Chloroquine as a Novel Therapeutic Strategy in Breast Cancer
Brief Title: A Phase 2 Randomized, Double-blind Trial Evaluating the Effects of Chloroquine in Breast Cancer
Acronym: CUBiC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OTT 14-02
Record Dates: First submitted 2015-01-05; First posted 2015-01-07 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer; Invasive Breast Cancer
Keywords: breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Chloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chloroquine (Experimental): The daily oral dose per patient is 500 mg of chloroquine. Patients may be taking the drug for 2-6 weeks leading up to the date of the surgery. The last dose will be taken the evening before surgery.
  Interventions: Drug: Chloroquine
- Placebo (Placebo Comparator): The daily oral dose per patient is 500 mg of placebo (lactose). Patients may be taking the drug for 2-6 weeks leading up to the date of the surgery. The last dose will be taken the evening before surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chloroquine — chloroquine 500 mg daily as an oral capsule during the wait time to surgery.
  Arms: Chloroquine
Drug: Placebo
  Arms: Placebo

SUMMARY:
Chloroquine (CQ) is a well known, well tolerated medication that has been used for many years traditionally for arthritis, lupus, and malaria. It has anti-inflammatory properties but is often the drug of choice for arthritis and malaria due to its few side effects. Recently, laboratory investigations have proven that CQ may potentially have anti-cancer properties, by inhibiting a process which allows cancers such as breast cancer to continue to grow (a process known as "autophagy"). Therefore, this study will look at how well CQ can inhibit the growth of breast cancers in patients while waiting for surgery.

DETAILED DESCRIPTION:
Patients diagnosed with breast cancer can sometimes wait up to 6 weeks for their surgery. The wait leading up to surgery is a potentially long and anxious time. Since no treatment is happening during this period anyway, this study will allow patients to receive CQ during this waiting period. This study will compare CQ treatment before surgery with the standard approach during this time, which is no treatment.

Although CQ is widely used for the treatment of arthritis and malaria, CQ is considered investigational for use in breast cancer.

The study will NOT interfere with the routine assessments as part of the pre-operative care, NOR will it delay the date of surgery.

This study compares the effects of the CQ to placebo. Participants will be randomized 1:1 and be provided with the blinded placebo or QC (500mg daily) during the wait time. Biomarker testing will be performed on the initial biopsy tissue and at the time of surgery as well as blood work. There is also an opportunity for participants to enrol in the optional sample collection for future research.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed histologically confirmed primary invasive breast cancer who is currently not undergoing any treatment while awaiting surgery in the next 2-6 weeks
* tumour ≥ 1.5 cm by palpation or imaging
* ECOG performance status 0-2
* written informed consent for the study

Exclusion Criteria:

* Known Metastatic breast cancer
* history of pre-existing known retinal or ocular pathology patient has only one functioning eye
* abnormal hepatic function (serum AST or ALT >3x upper limit of normal)
* currently on CQ or HCQ or has been on the drug within the past 3 months for other conditions
* known history of psoriasis
* known history of epilepsy or seizures
* electrocardiogram showing QT prolongation based on QTc interval >450 ms
* inability to comply with a study protocol (abuse of alcohol, drugs or psychotic states)
* current known pregnancy or actively nursing
* allergic reactions to quinolones or CQ
* inability to consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Effect of a brief course of CQ on tumour proliferation and apoptosis | baseline and at 2-6 weeks, the day of surgery
  We will assess relative changes in proliferative and apoptotic response indices based on Ki67 and TUNEL assays in primary breast cancer biopsies pre- and post-treatment with CQ, as these changes occur more rapidly than gross changes in tumour volume.

SECONDARY OUTCOMES:
Measure of Circulating CQ Metabolites | baseline and at 2-6 weeks, the day of surgery
  Plasma samples collected at baseline and at surgery will be assessed for levels of CQ and its metabolite desethylchloroquine (DECQ) by high-performance liquid chromatography (HPLC) as described
Autophagic Markers in Cancerous and Stromal Tissue | baseline and at 2-6 weeks, the day of surgery
  Immunohistochemical detection of proteins such as Beclin 1, LC3, and p62 which are required for autophagosome formation have been extensively studied in clinical tumour samples, and will be assessed in participant samples pre and post-CQ treatment.

OTHER OUTCOMES:
Assessment of Toxicity of CQ in Breast Cancer Patients | baseline and at 2-6 weeks, the day of surgery
  Even through CQ has an excellent safety profile and the dose of 500 mg/day is well within the dosage in which toxicity is measured, all adverse and serious adverse events while on CQ will be monitored as per the study assessments calendar via the Health Canada Pharmacovigilance program, Ottawa Hospital Science Network-REB and Data Safety Monitoring Board. As the most serious adverse events with CQ use are ocular events, the American Academy of Ophthalmology recommends ophthalmologic screening and management of patients on CQ. Given the limited duration patients will be taking CQ, it is not expected that any ocular events will be observed, however, for enhanced safety, we have 3 ophthalmology collaborators and we will mandate intense vigilance with an ophthalmologic screening exam at baseline, at one month post surgery, and a final at 4-6 months after stopping CQ.
Differential Gene and Expression using Microarray Analysis. | baseline and at 2-6 weeks, the day of surgery
  The breast cancer tissue collected and stored during this clinical trial will offer a unique opportunity to study the effect of CQ on the biology of human breast tissue. RNA and gene expression levels will be extracted from participant samples that have been treated with CQ. Potential differentially expressed targets will be confirmed by quantitative RT-PCR using specific primers and normalization to endogenous β-actin or GAPDH as controls.

CONTACTS AND LOCATIONS:
Overall Officials: Angel Arnaout, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital Woman's Breast Health Centre, Ottawa, Ontario, Canada